CLINICAL TRIAL: NCT06717490
Title: Effect of Magnesium Sulfate on Postoperative Hypercoagulability Using Thromboelastometry in Laparoscopic Gynecological Surgeries
Brief Title: Magnesium Sulfate and Postoperative Hypercoagulability in Laparoscopic Gynecological Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marianna Mavromati (Other)
Collaborators: Aretaieion University Hospital (Other)
Responsible Party: Sponsor-Investigator, Marianna Mavromati, Marianna Mavromati, MD, Principal Investigator and Anesthesiology Resident, Aretaieion University Hospital, NKUA, Aretaieion University Hospital
Organization: Aretaieion University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 619/05-11-2024
Record Dates: First submitted 2024-11-20; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Magnesium Sulfate; Thromboelastometry
MeSH Terms: interventions — Magnesium Sulfate; Thrombelastography

STUDY DESIGN:
Intervention Model Description: Patients are divided into two groups, with one group receiving magnesium sulfate and the other receiving normal saline.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MS group (Active Comparator): The patients allocated to this group will receive an intravenous bolus of magnesium sulfate (50 mg/kg) followed by a continuous infusion (15 mg/kg/h) Blood coagulation parameters will be assessed pre- and post- magnesium administration using thromboelastometry.
  Interventions: Drug: Magnesium sulphate
- NS group (Placebo Comparator): The patients allocated to this group will receive an equivalent volume of normal saline proportionally to the active comparator group. Blood coagulation parameters will be assessed pre- and post-magnesium administration using thromboelastometry.
  Interventions: Other: Placebo Drug

INTERVENTIONS:
Drug: Magnesium sulphate — In patients allocated to the MS group, a fixed dose of magnesium sulfate diluted in a fixed volume of natural saline will be administered intravenously.
  Thromboelastometry will be performed pre and post magnesium administration.
  Other Names: Thromboelastometry
  Arms: MS group
Other: Placebo Drug — In patients allocated to the NS group, a fixed dose of natural saline will be administered intravenously, through a fixed volume of solution.
  Thromboelastometry will be performed pre and post magnesium administration.
  Other Names: Thromboelastometry
  Arms: NS group

SUMMARY:
This will be a prospective randomized, double-blind study, aiming at investigating the effects of magnesium sulfate on postoperative hypercoagulability in patients undergoing laparoscopic gynecological surgeries under general anesthesia

DETAILED DESCRIPTION:
This randomized, double-blind, controlled study investigates the effects of magnesium sulfate on postoperative hypercoagulability in patients undergoing laparoscopic gynecological surgeries under general anesthesia. Using thromboelastometry, the study aims to assess the impact of magnesium sulfate on blood coagulation parameters. Patients are divided into two groups, with one group receiving magnesium sulfate and the other receiving normal saline. Both patients and investigators are blinded to the treatment allocation. The study will analyze clotting time, clot formation, and coagulation markers to evaluate the therapeutic potential of magnesium sulfate in reducing postoperative hypercoagulability.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients
* Laparoscopic gynecological surgeries
* age >18 years
* Patients receiving prophylactic anticoagulant therapy 12 hours before surgery based on the Caprini score
* Patients receiving prophylactic anticoagulant therapy 12 hours postoperatively based on the Caprini score.

Exclusion Criteria:

* ASA ≥ III
* age <18 years
* BMI >40 kg/m²
* Pregnancy
* Known hematologic disorders
* Liver/kidney/cardiovascular disease
* Severe anemia (6,5- 7,9 g/dl)
* Inability or refusal to provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants include individuals with biologically female internal reproductive organs (e.g., XX chromosomes and uterus), regardless of their self-identified gender.
Enrollment: 60 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Clotting Time [CT] (in seconds, measured using ROTEM) | Up to six hours (first thromboelastometry will be performed immediately before magnesium administration intraoperatively, and the second thromboelastometry will be performed at the post-anesthesia care unit)
  Clotting Time [CT] is measured using Thromboelastometry (ROTEM) as part of coagulation parameters. CT represents the time (in seconds) required for the initial clot formation in the blood sample
Clot Formation Time [CFT] (in seconds, measured using ROTEM) | Up to six hours (first thromboelastometry will be performed immediately before magnesium administration intraoperatively, and the second thromboelastometry will be performed at the post-anesthesia care unit)
  Clot Formation Time [CFT] is measured using Thromboelastometry (ROTEM) to evaluate the time required for the clot to stabilize. CFT is expressed in seconds and represents the time to achieve adequate clot firmness in the blood sample
Maximum Clot Firmness [MCF] (in mm, measured using ROTEM) | Up to six hours (first thromboelastometry will be performed immediately before magnesium administration intraoperatively, and the second thromboelastometry will be performed at the post-anesthesia care unit)
  Maximum Clot Firmness [MCF] is measured using Thromboelastometry (ROTEM) to evaluate the maximum stability of the clot. MCF is expressed in millimeters and represents the highest clot firmness achieved in the blood sample
a-angle (in degrees, measured using ROTEM) | Up to six hours (first thromboelastometry will be performed immediately before magnesium administration intraoperatively, and the second thromboelastometry will be performed at the post-anesthesia care unit)
  a-angle measured using Thromboelastometry (ROTEM) to assess the rate of fibrin polymerization and clot formation dynamics. The a-angle is expressed in degrees (°) and indicates the speed of fibrin build-up

SECONDARY OUTCOMES:
Train of Four (TOF) | 4 minutes (time point 0 will be at neuromuscular blocking agent administration)
  Train of Four (TOF) will be measured using a neuromuscular stimulator to assess neuromuscular blockade. Measurements will be noted at the induction of general anesthesia after neuromuscular blocking agent administration until TOF reaches zero
Area Under the Curve (AUC) for Nociception Index Level (NOL) | Intraoperative
  Nociception Index Level (NOL) will be measured using the NOL monitoring system. Measurements will be performed throughout the surgery, and the area under the curve (AUC) will be calculated to evaluate nociceptive responses.
Changes in INR Before and After Magnesium Administration | Up to six hours (first assessment will be performed before surgery and the second assessment will be performed at the post-anesthesia care unit)
  Changes in INR (International Normalized Ratio) will be assessed before and after magnesium administration using an automated coagulation analysis system
Changes in aPTT Before and After Magnesium Administration | Up to six hours (first assessment will be performed before surgery and the second assessment will be performed at the post-anesthesia care unit)
  Changes in aPTT will be assessed before and after magnesium administration using an automated coagulation analysis system
Changes in PT Before and After Magnesium Administration | Up to six hours (first assessment will be performed before surgery and the second assessment will be performed at the post-anesthesia care unit)
  Changes in platelet count will be assessed before and after magnesium administration using a hematology analyzer
Changes in Platelet Count Before and After Magnesium Administration | Up to six hours (first assessment will be performed before surgery and the second assessment will be performed at the post-anesthesia care unit)
  Changes in platelet count will be assessed before and after magnesium administration using a hematology analyzer
Changes in Fibrinogen Levels Before and After Magnesium Administration | Up to six hours (first assessment will be performed before surgery and the second assessment will be performed at the post-anesthesia care unit)
  Changes in fibrinogen levels will be assessed before and after magnesium administration using the Clauss method
Clinical thrombosis symptoms | 24 hours (first assessment will be performed immediately before surgery, and the final assessment will be performed 24 hours postoperatively)
  Symptoms of clinical thrombosis (e.g., redness, swelling, pain) will be assessed through physical examination by the attending physician before and after magnesium administration

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, Professor, Study Chair — Aretaieio University Hospital, National and Kapodistrian University of Athens
Locations (1):
- Aretaieion University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No